CLINICAL TRIAL: NCT07260656
Title: A Double-Blind, Randomized, Pilot Study to Investigate the Efficacy of a Topical Palmitated Formulation of Capsaicin (Capsadyn®) In the Treatment of Diabetic Neuropathic Foot Pain
Brief Title: Efficacy of a Topical Palmitated Formulation of Capsaicin (Capsadyn®) In the Treatment of Diabetic Neuropathic Foot Pain
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-25-2072
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Neuropathies, Painful; Diabetic Foot; Diabetic Peripheral Neuropathy
Keywords: diabetic foot pain
MeSH Terms: conditions — Diabetic Neuropathies; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The participant population will be scheduled for an even split between the two study arms.
Who Masked: Participant, Investigator
Masking Description: Pharmacist will randomize participants 1:1 between the two arms, either Capsadyn or placebo. Study products will provide blinded product to study staff to provide to participants in coded, white-labeled, one ounce plastic jars.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Capsadyn Arm (Active Comparator): participant will receive an over-the-counter topical cream with .25% capsaicin palmitate
  Interventions: Drug: Capsaicin Palmitate
- Placebo Arm (Placebo Comparator): participant will receive an over-the counter topical cream with no active ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capsaicin Palmitate — Participant will apply a small amount of topical cream (size of a quarter) to one or both feet twice a day, once in the morning and once in the evening.
  Other Names: Capsadyn
  Arms: Capsadyn Arm
Drug: Placebo — Participant will apply a small amount of topical cream (size of a quarter) to one or both feet twice a day, once in the morning and once in the evening.
  Other Names: OTC topical cream
  Arms: Placebo Arm

SUMMARY:
The purpose of this research is to assess whether the use of a topical cream with an active ingredient can reduce the amount of foot pain experienced in participants who have been diagnosed with Diabetic Peripheral Neuropathy (DPN) with minimal side effects or discomfort from use.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled trial with two arms to assess the pain-reducing effects of topical Capsadyn compared to a placebo (carrier cream). At the appointment/recruitment visit, patients will receive standard of care as determined by their clinician. At the first visit, participants opting into the trial will not receive any new medications designed for producing pain relief alongside the Test Article but will continue medications taken before entry to the study, if use history is stable, or medications not specifically designed for pain reduction. Both the clinician administering the Test Article and the participant will be blinded to Test Article, or unaware of whether it is Capsadyn or placebo.

A Test article can be administered to either a unilateral area, or bilateral painful areas. Test Article should be administered over the complete painful area. Test Articles will be packaged in coded, white-labeled one-ounce plastic jars, marked only with a code indicating Capsadyn or placebo, and sent to Carilion Pharmacy for distribution to healthcare providers. The pharmacy will quarantine the Test Articles and randomize Test Article scheduling between the two arms. The participant population will be scheduled for an even split between the two study arms. With the recruitment of 40 participants (20 per group), an interim look at the data will be done to assess participant compliance with instructions, general progress of the study and to troubleshoot any issues that may have arisen.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 toes per foot
* Have otherwise intact feet.
* Absence of any eczema, hyperkeratosis, scleroderma, or other dermatological conditions afflicting the area of Test Article administration that may interfere with absorption, particularly hyperhidrosis.
* Must agree to apply the Test Article to painful areas of feet as directed by research personnel.
* Must agree to apply the Test Article to feet as instructed 2x per day.
* Must wait 60 minutes after each application of Test Article before filling out NRS forms.
* Unless burning is encountered soon after application, the participant must wait at least 60 minutes before washing feet after application of Test Article.
* All participants must be willing to use Test Articles blinded.

Exclusion Criteria:

* Younger than 25 and older than 75 years of age
* Any dermatological condition(s) with the potential to disrupt skin integrity or alter sensory function of the feet.
* Any open wounds, skin ulceration, infection, skin irritation (e.g., poison oak), history of eczema, trauma or burn (including sunburn) affecting the feet within 30 days.
* Any recent medical history of surgery affecting the feet.
* Unless part of a stable continuum of substance use prior to start of study, the use of any topical medication products on feet, including holistic formulations, patch or herbal products, cannabinoid products, prescription or over the-counter (OTC) analgesic creams/lotions/patches/gels, nonsteroidal anti-inflammatory drugs, acetaminophen, counterirritants, local anesthetics, or steroids is prohibited.
* Current substance abuse.
* History of hypersensitivity or allergy to chili peppers, coconut oil, Shea butter, or sunflower seed oil.
* Except for interventions for mobility, (e.g., physical therapy, exercise, grounding) no concurrent foot therapy for pain that may interfere with NRS evaluations is permitted (e.g., massage, electrophoresis, red light, etc.).
* No concurrent enrollment in another clinical trial.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Significant reduction in foot pain in participants with chronic diabetic neuropathic foot pain. | A NRS will be completed by the participant twice a day, once in the morning and once in the evening, for 14 days after each application of the topical cream provided
  Participants will complete a Numeric Rating Scale (NRS) twice a day for 14 days one hour after applying topical cream to the area of their foot where they are experiencing Diabetic Peripheral Neuropathy foot pain. Participants will not be aware of whether the topical cream applied includes capsaicin palmitate. The NRS rates the intensity of symptoms with a scale of 0 to 10 with 0 being no symptom present to 10 being the worst possible intensity. The symptoms being assessed include redness, irritation, itching, tingling, and a burning or cooling sensation one hour after applying the topical cream.
  Study investigators will review the variances in the NRS ratings throughout the duration of the 14 days of all participants and report any changes from baseline scores. Data will be analyzed using one-way repeated measures ANOVA, followed by the Mann-Whitney U post-hoc test. Data will be visualized as box-and-whisker plots, comparing Capsadyn to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Carpenter, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No